CLINICAL TRIAL: NCT05814796
Title: Assessment of Obstructive Sleep Apnea Syndrome in Non-Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Atef Mohammed MohammedElgalaly, Resident doctor, Assiut University
Other Study IDs: sleep apnea in non obese
Record Dates: First submitted 2023-01-18; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients: BMI>30
- Non obese: Overweight: BMI = 25-29.9 Normal weight: BMI = 18.5-24.9

SUMMARY:
The aim of this study is to evaluate OSAS in non-obese patients, and to compare patient characteristics, clinical markers between obese and non-obese patients.

DETAILED DESCRIPTION:
OSAS (obstructive sleep apnea syndrome) is characterized by repeated collapses of the upper airways that result in a marked reduction (hypopnea) or complete interruption (apnea) of the airflow. Polysomnography is the gold standard tool for diagnosis. OSAS is defined broadly as an apnea-hypopnea index (AHI) greater than five events per hour of sleep.

The events of apneas and hypopneas are followed by phasic oxyhemoglobin desaturations, with consequent intermittent hypoxemia, sympathetic hyperactivation, and sleep fragmentation. This results in many complications such as: atherosclerosis, acute coronary syndrome , diabetes , stroke , premature death , reduction of cognitive functions and quality of life .

OSA is the most common sleep-related breathing disorder (SRBD). The estimated prevalence in North America is approximately 15- 30 % in males and 10 - 15 % in females . Global estimates using five or more events per hour suggest rates of 936 million people worldwide with mild to severe OSAS, and 425 million people worldwide with moderate to severe OSAS, between the ages of 30 and 69 years of age . OSA has a racial predisposition. It is more prevalent in African Americans who are younger than 35 years old compared with White Americans of the same age group, independent of body weight . The prevalence of OSAS appears to be increasing and may be related to the increasing rates of obesity and increased detection rates of OSA .

It is well known that obesity is the main risk factor for OSAS . On the other hand, there are multiple risk factors than can occur in non-obese. These risk factors include anatomical factors e.g. retrognathia, soft palate laxity, craniofacial conformations of reduced dimensions and macroglossia, which lead to greater collapse of the upper airways in non-obese patients . In addition, genetic predisposition, smoking, alcohol consumption, and gender play a role as risk factors for OSAS. The different pathophysiological mechanisms results in different disease phenotypes .

Pathophysiology of OSAS is complex. This include: instability of ventilatory control, also known as high loop gain, neuromuscular inefficiency of the dilator muscles of the upper airways and reduced awakening threshold, also known as low arousal threshold The relation of obesity with OSAS is well-established, and has been thoroughly investigated. However, the proportion of patients with OSAS who are not obese, their clinical presentation, pathophysiological mechanisms and response to therapies has been minimally investigated .

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 yrs. old. 2.Informed consent to participate in the study is provided.

   Exclusion Criteria:
   * 1. Pregnancy
2. Neuromuscular disorders
3. Psychiatric instability
4. Suspected narcolepsy
5. Uncontrolled cardiovascular disease (uncontrolled hypertension, heart failure, uncontrolled arrhythmia)
6. Cheynes-Stokes syndrome
7. Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients addmitted to Chest Department, Assuit University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
evaluate OSAS in non-obese patients, and to compare patient characteristics, clinical markers between obese and non-obese patients. | basline
  Weight in kilograms and height in meters weight and height will be combined to report BMI in kg/m^2).